CLINICAL TRIAL: NCT00430183
Title: A Randomized Phase III Study of Neo-Adjuvant Docetaxel and Androgen Deprivation Prior to Radical Prostatectomy Versus Immediate Radical Prostatectomy in Patients With High-Risk, Clinically Localized Prostate Cancer
Brief Title: Surgery With or Without Docetaxel and Leuprolide or Goserelin in Treating Patients With High-Risk Localized Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB 90203; U10CA031946 (NIH); CDR0000526353 (Other: Physician Data Query)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Gonadotropin-Releasing Hormone; Leuprolide; Goserelin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: docetaxel + LHRH agonist + surgical intervention (Experimental): Patients receive six cycles of docetaxel administered every 3 weeks combined with 18-24 weeks of androgen deprivation therapy. During each cycle of chemotherapy, all patients should undergo premedication with dexamethasone 8 mg orally prior to docetaxel. Dexamethasone may also be given intravenously according to institutional guidelines.
  Patients will also receive androgen deprivation for 18-24 weeks of an LHRH agonist (eg, leuprolide acetate, goserelin acetate). Additional premedication and antiemetics may be given at the physician's discretion and as defined by the protocol.
  Patients will undergo standard surgical intervention. The surgical procedures will be performed within 60 days of the completion of neoadjuvant therapy. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. It must be initiated within 6 months of the date of surgery.
  Interventions: Drug: docetaxel; Drug: LHRH agonist; Procedure: surgery
- Arm B: surgical intervention (Other): All patients undergo standard surgical intervention. The surgical procedures will be performed within 60 days of randomization. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. Adjuvant radiation must be initiated within 6 months of the date of surgery.
  Interventions: Procedure: surgery

INTERVENTIONS:
Drug: docetaxel — 75 mg/m^2 will be administered intravenously over one hour on Day 1 of each cycle, every 21 days
  Arms: Arm A: docetaxel + LHRH agonist + surgical intervention
Drug: LHRH agonist — Given intramuscularly
  Other Names: leuprolide acetate OR; goserelin acetate
  Arms: Arm A: docetaxel + LHRH agonist + surgical intervention
Procedure: surgery — Patients undergo radical prostatectomy with staging pelvic lymphadenectomy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as goserelin and leuprolide, may stop the adrenal glands from making androgens. Giving docetaxel and leuprolide or goserelin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether giving docetaxel and leuprolide or goserelin before surgery is more effective than surgery alone in treating patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying docetaxel and leuprolide or goserelin to see how well they work when given before surgery compared with surgery alone in treating patients with high-risk localized prostate cancer.

DETAILED DESCRIPTION:
This randomized trial tests whether the addition of chemohormonal therapy improves PSA-progression free survival in patients with high risk, clinically-localized prostate cancer. The neoadjuvant approach is taken since there appears to be a higher acceptance rate in the prostate population for this type of therapy and several phase II trials have demonstrated its safety. Multiple chemotherapeutic therapies have shown efficacy in advanced prostate cancer and docetaxel has become the community standard. Many high risk patients are initiated on LHRH agonists at or near the time of diagnosis of their prostate cancer. In order to allow the inclusion of these patients in the protocol, enhanced enrollment and maintain compliance with therapy, up to 3 months of androgen deprivation therapy prior to enrollment will be permitted. This study will therefore be able to test the hypothesis that targeting both androgen-sensitive and chemotherapy- sensitive prostate cancer cells will improve outcomes in these high-risk patients.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to nomogram-predicted biochemical progression-free survival at 5 years (0-20.9% vs 21-39.9% vs 40-59.9% vs ≥ 60%) and androgen-deprivation therapy prior to randomization ≤ 4 months (no vs yes). Patients are randomized to 1 of 2 treatment arms. Please see the Arms sections for more details.

The primary and secondary objectives are described below.

Primary:

- To determine whether treatment with neoadjuvant docetaxel and androgen deprivation therapy prior to radical prostatectomy will increase the rate of 3-year biochemical progression-free survival (bPFS) compared to treatment with immediate radical prostatectomy alone for high-risk prostate cancer patients.

Secondary:

* To compare the 5-year bPFS rate, bPFS, disease progression, disease-free survival, and overall survival of patients randomized to the two arms of this trial
* To determine the safety and tolerability of neoadjuvant docetaxel and androgen deprivation therapy prior to surgery for high-risk patients undergoing radical prostatectomy
* To compare the impact of neoadjuvant docetaxel and androgen deprivation therapy on time to clinically apparent local disease recurrence and metastatic disease in high-risk patients undergoing radical prostatectomy for clinically localized prostate cancer
* To compare the impact of neoadjuvant docetaxel and androgen deprivation therapy relative to RP on pathologic tumor stage, frequency of lymph node metastases and positive margin rates for high-risk patients undergoing radical prostatectomy for clinically localized prostate cancer
* To determine if changes in serum testosterone levels will predict bPFS
* To determine prospectively whether PSA doubling time (PSADT) is a surrogate endpoint for time to clinical metastases and overall survival

Patients are followed up to 15 years post-randomization.

ELIGIBILITY:
1. Histologic documentation - Histologic documentation of prostatic adenocarcinoma.

   Patients with small cell, neuroendocrine, or transitional cell carcinomas are not eligible.

   All eligible patients must have a known Gleason sum based on biopsy or TURP at the time of registration.
2. Clinically localized disease - Patients must have clinical stage T1-T3a and no radiographic evidence of metastatic disease as demonstrated by:

   * EITHER CT or MRI of the abdomen and pelvis, OR endorectal MRI of the pelvis that demonstrate no nodes > 1.5 cm. If one or more pelvic lymph node(s) measures > 1.5 cm, a negative biopsy is required. If more than one lymph node is > 1.5 cm, the largest or most accessible node should be biopsied.

   AND
   * Negative bone scan (with plain films and/or MRI and/or CT scan confirmation, if necessary). Positive PET and Prostascint scans are not considered proof of metastatic disease.
3. Determination of high-risk status: Patients must have either:

   * A Kattan nomogram predicted probability of being free from biochemical progression at 5 years after surgery of < 60%.

   OR
   * Prostate biopsy Gleason sum ≥ 8 (NOTE: The Kattan nomogram probability must be calculated for all patients, including those eligible based on Gleason sum ≥ 8 only.)
4. Prior treatment - No prior treatment for prostate cancer including prior surgery (excluding TURP), pelvic lymph node dissection, radiation therapy, or chemotherapy.

   Patients may have received up to 4 months of androgen deprivation therapy (LHRH agonists, antiandrogens, or both) prior to being enrolled on the study.
5. Appropriate surgical candidates - Patients must be appropriate candidates for radical prostatectomy with an estimated life expectancy > 10 years as determined by a urologist. Evidence of underlying cardiac disease should be evaluated prior to enrollment to ensure that patients are not at high risk of cardiac complications.
6. Clotting history - Patients with a history of deep venous thrombosis, pulmonary embolism, and/or cerebrovascular accident or currently requiring systemic anticoagulation are eligible provided they are determined to be candidates for radical prostatectomy.
7. ECOG performance status: 0-2
8. Age: ≥ 18 years of age
9. Required Initial Laboratory Values:

   * ANC ≥ 1500/μL
   * Platelet count ≥ 150,000/μL
   * Creatinine ≤ 2.0 mg/dL
   * Pre-registration serum PSA level ≤ 100 ng/mL
   * Bilirubin ≤ 1.5XULN (2.5XULN in patients with Gilbert's disease)
   * AST/ALT ≤1.5XULN

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2007-05-08 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2030-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (226):
- United States (221):
  - Providence Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - University of California Davis Cancer Center, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - California Pacific Medical Center - Pacific Campus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center, Vallejo, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Veterans Affairs Medical Center - West Haven, West Haven, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Delnor Hospital - Geneva, Geneva, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - St. Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Tufts Medical Center Cancer Center, Boston, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Healthcare - Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Carolinas Medical Center - Union, Monroe, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Regional Medical Center, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (5):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec

REFERENCES:
- [Derived] Eastham JA, Heller G, Halabi S, Monk JP 3rd, Beltran H, Gleave M, Evans CP, Clinton SK, Szmulewitz RZ, Coleman J, Hillman DW, Watt CR, George S, Sanda MG, Hahn OM, Taplin ME, Parsons JK, Mohler JL, Small EJ, Morris MJ. Cancer and Leukemia Group B 90203 (Alliance): Radical Prostatectomy With or Without Neoadjuvant Chemohormonal Therapy in Localized, High-Risk Prostate Cancer. J Clin Oncol. 2020 Sep 10;38(26):3042-3050. doi: 10.1200/JCO.20.00315. Epub 2020 Jul 24. PMID 32706639
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Docetaxel + LHRH Agonist + Surgical Intervention: Patients receive six cycles of 75 mg/m^2 docetaxel administered every 3 weeks combined with 18-24 weeks of androgen deprivation therapy. During each cycle of chemotherapy, all patients should undergo premedication with dexamethasone 8 mg orally prior to docetaxel. Dexamethasone may also be given intravenously according to institutional guidelines.Patients will also receive androgen deprivation for 18-24 weeks of an LHRH agonist (eg, leuprolide acetate, goserelin acetate). Additional premedication and antiemetics may be given at the physician's discretion and as defined by the protocol. Patients will undergo standard surgical intervention. The surgical procedures will be performed within 60 days of the completion of neoadjuvant therapy. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. It must be initiated within 6 months of the date of surgery.
- Arm B: Surgical Intervention: All patients undergo standard surgical intervention. The surgical procedures will be performed within 60 days of randomization. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. Adjuvant radiation must be initiated within 6 months of the date of surgery(surgery: Patients undergo radical prostatectomy with staging pelvic lymphadenectomy).
Period: Overall Study
Arm/Group | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention | Arm B: Surgical Intervention
Started | 391 | 397
Completed | 391 | 397
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Docetaxel + LHRH Agonist + Surgical Intervention: Patients receive six cycles of 75 mg/m^2 docetaxel administered every 3 weeks combined with 18-24 weeks of androgen deprivation therapy. During each cycle of chemotherapy, all patients should undergo premedication with dexamethasone 8 mg orally prior to docetaxel. Dexamethasone may also be given intravenously according to institutional guidelines.> > Patients will also receive androgen deprivation for 18-24 weeks of an LHRH agonist (eg, leuprolide acetate, goserelin acetate). Additional premedication and antiemetics may be given at the physician's discretion and as defined by the protocol. >
  > Patients will undergo standard surgical intervention. The surgical procedures will be performed within 60 days of the completion of neoadjuvant therapy. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. It must be initiated within 6 months of the date of surgery.
- Arm B: Surgical Intervention: All patients undergo standard surgical intervention. The surgical procedures will be performed within 60 days of randomization. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. Adjuvant radiation must be initiated within 6 months of the date of surgery (surgery: Patients undergo radical prostatectomy with staging pelvic lymphadenectomy).
- Total: Total of all reporting groups
Arm/Group | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention | Arm B: Surgical Intervention | Total
Number analyzed (Participants) | 391 | 397 | 788
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 78] | 63 [33 to 84] | 63 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 391 | 397 | 788
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 330 | 337 | 667
  Race: Black | 40 | 38 | 78
  Race: Other | 15 | 9 | 24
  Race: Unknown | 6 | 13 | 19
Clinical stage by digital rectal examination (Primary Tumor (T) Stage) [Count of Participants; unit: Participants] — The stage of cancer (amount or spread of cancer in the body) that is based on digital rectal examination performed prior to surgery. The primary tumor (T) stage using the TNM system is reported here. TX: Main tumor cannot be measured.>> T0: Main tumor cannot be found.>> T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 102 | 129 | 231
    T2 | 219 | 204 | 423
    T3a | 70 | 64 | 134

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Biochemical Progression-Free Survival (bPFS Proportion) at 3 Years
Description: Proportion of participants surviving 3 years from randomization without biochemical progression or death. bPFS was defined as the time from randomization to the date of the first documented biochemical progression or death. Progression will be defined as having experienced either of the following: a serum PSA level > 0.2 ng/mL that increases on 2 consecutive occasions each of which is at least 3 months apart or death occurs. The time of biochemical failure is measured from the date of randomization to the date of the first PSA level > 0.2 ng/mL.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention | Arm B: Surgical Intervention
Number analyzed (Participants) | 391 | 397
proportion of patients | 0.89 [0.87 to 0.91] | 0.84 [0.78 to 0.90]

2. Secondary Outcome: 5-year bPFS Rate
Description: Proportion of participants surviving 5 years from randomization without biochemical progression or death.
Time Frame: 5 years
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention | Arm B: Surgical Intervention
Number analyzed (Participants) | 391 | 397
Proportion of participants | 0.81 | 0.74

3. Secondary Outcome: Time to Clinical Local Recurrence (The Time From Randomization to the First Biopsy-proven Recurrence in the Prostatic Bed or New Mass.)
Time Frame: Up to 15 years post-randomization
Reporting Status: Not Posted, anticipated posting 2030-10

4. Secondary Outcome: Time to Metastatic Disease Progression (The Date of Randomization to Date of Evidence of Systemic Disease on Bone Scan or Cross Sectional Imaging.)
Time Frame: Up to 15 years post-randomization
Reporting Status: Not Posted, anticipated posting 2030-10

5. Secondary Outcome: Unacceptable Toxicity (Grade 3 or Higher Toxicity)
Time Frame: Up to 15 years post-randomization
Reporting Status: Not Posted, anticipated posting 2030-10

6. Secondary Outcome: Prostate Cancer-specific-free Survival (The Time From Randomization to the Time of Death Due to Prostate Cancer.)
Time Frame: Up to 15 years post-randomization
Reporting Status: Not Posted, anticipated posting 2030-10

7. Secondary Outcome: Disease Progression
Time Frame: Up to 15 years post-randomization
Reporting Status: Not Posted, anticipated posting 2030-10

8. Secondary Outcome: Overall Survival (The Date of Randomization to the Time of Death Due to Prostate Cancer.)
Time Frame: Up to 15 years post-randomization
Reporting Status: Not Posted, anticipated posting 2030-10

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Per protocol, only Arm A patients were assessed for adverse events (i.e. Serious, and Other (Not Including Serious) Adverse Events). All-Cause Mortality is monitored for all patients.
Groups:
- Arm A: Docetaxel + LHRH Agonist + Surgical Intervention: Patients will undergo standard surgical intervention. The surgical procedures will be performed within 60 days of the completion of neoadjuvant therapy. Patients are allowed to receive adjuvant external beam radiation at the discretion of the treating physician and as defined per the protocol. It must be initiated within 6 months of the date of surgery.
Arm/Group | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention | Arm B: Surgical Intervention
All-Cause Mortality (participants affected / at risk) | 39/391 | 54/397
Serious Adverse Events (participants affected / at risk) | 31/391 | 0/0
Other Adverse Events (participants affected / at risk) | 361/391 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention (N=391) | Arm B: Surgical Intervention (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (8) | 0 (0)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (14) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Edema limbs (General disorders) | 4 (5) | 0 (0)
Fatigue (General disorders) | 20 (26) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (4) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (11) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (9) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (9) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Docetaxel + LHRH Agonist + Surgical Intervention (N=391) | Arm B: Surgical Intervention (N=0)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (14) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 128 (255) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 102 (221) | 0 (0)
Nausea (Gastrointestinal disorders) | 158 (380) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 42 (67) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 116 (249) | 0 (0)
Fatigue (General disorders) | 322 (1340) | 0 (0)
Fever (General disorders) | 2 (3) | 0 (0)
Localized edema (General disorders) | 6 (8) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 54 (84) | 0 (0)
Bladder infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 5 (6) | 0 (0)
Tooth infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Intraop. inj. - NERVE: facial sens-taste (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 10 (13) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 19 (29) | 0 (0)
Lymphocyte count decreased (Investigations) | 15 (19) | 0 (0)
Neutrophil count decreased (Investigations) | 96 (173) | 0 (0)
Platelet count decreased (Investigations) | 12 (17) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 25 (55) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (6) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 126 (306) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 152 (400) | 0 (0)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (5) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (5) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 188 (512) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (8) | 0 (0)
Depression (Psychiatric disorders) | 3 (8) | 0 (0)
Euphoria (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (19) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (7) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 6 (17) | 0 (0)
Feminization (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pharyngeal mucositis (funct/sympt) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (16) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 108 (217) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 11 (23) | 0 (0)
Hypertension (Vascular disorders) | 7 (19) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Vascular disorder (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT00430183/Prot_SAP_000.pdf